CLINICAL TRIAL: NCT03522324
Title: An Observational Study of the Effects of Edible Cannabis and Its Constituent Cannabinoids on Pain, Inflammation, and Cognition
Brief Title: Pain Research: Innovative Strategies With Marijuana
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other); Colorado State University (Other)
Responsible Party: Principal Investigator, L. Cinnamon Bidwell, Assistant Research Professor, University of Colorado, Boulder
Other Study IDs: R01AT009541 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-05-11 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Chronic Low Back Pain; Cannabis Use
Keywords: Cannabis; Pain; Cytokines; Inflammation; Cognition
MeSH Terms: conditions — Chronic Pain; Marijuana Abuse; Pain; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples collected for cytokine and cannabinoid quantitation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cannabis Edible — Self-Directed Use (ad-libitum)

SUMMARY:
This study tests the effects of cannabinoid levels in blood on pain relief, inflammation, and cognitive dysfunction in chronic pain patients who choose to use edible cannabis. Over a two-week period, participants use an edible product of their choice. Blood levels of 9-delta-tetrahydrocannabinol (THC) and cannabidiol (CBD) will be measured before, during, and after the two-week exposure period to determine whether there are associations with pain, inflammation, sleep, physical activity, anxiety/depression, and cognitive dysfunction. After the two-week self-administration period, participants will be followed for six months to collect self-report data on cannabis use, pain levels, sleep quality, and mental health symptoms.

DETAILED DESCRIPTION:
The National Center for Health Statistics reports that approximately 76 million Americans suffer from chronic pain, affecting the lives of more Americans than cancer, diabetes, and heart disease combined. Perhaps because of its ubiquity and the challenge to its treatment, relief from chronic pain is by far the most commonly cited condition by patients for use of marijuana, with 87%-94% of medical marijuana users reporting using for relief of a pain condition.

Although the mechanisms are still unclear, marijuana and its constituent cannabinoids, including 9-delta-tetrahydrocannabinol (THC), are thought to be involved in reducing pain and associated inflammation. However, THC is also associated with harm in the form of cognitive dysfunction. Synergistic interactions of multiple cannabinoids are believed to produce different effects on both pain relief and cognitive function as compared to THC alone. For example, cannabidiol (CBD) is another primary cannabinoid that may work synergistically with THC in a multi-target analgesic approach.

This study examines the effects of cannabinoids in edible form on pain relief, inflammation, and cognitive dysfunction in chronic pain patients who choose to use marijuana in the context of a short-term (2 weeks), patient-oriented, observational design and a mobile pharmacology and phlebotomy lab.

ELIGIBILITY:
Inclusion Criteria:

* Intent to initiate use of marijuana to treat chronic pain
* At least one episode of lifetime marijuana use, but infrequent marijuana use for prior six months
* Self-reported non-specific chronic low back pain for at least three months
* Health eligibility approved by study physician
* At least mild to moderate pain intensity OR pain interferes with important life functions

Exclusion Criteria:

* Other drug use (cocaine, methamphetamine, etc.) in the past 3 days and/or actively seeking or in treatment for any substance use disorder
* Use of marijuana to treat pain at any time in lives
* Current use of psychotropic medications (other than SSRIs and ADHD meds), or use of antivirals, steroids, or regular use of maximal doses of NSAIDS
* A daily tobacco user
* Are currently pregnant or trying to become pregnant
* Acute illness (other than chronic pain) or any immune-related disease (e.g., HIV)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cinnamon Bidwell, PhD, Principal Investigator — Institute of Cognitive Science, University of Colorado, Boulder
Locations (1):
- Center for Innovation and Creativity, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Melendez SN, Ortiz Torres M, Lisano JK, Giordano G, Skrzynski C, Hutchison KE, Bryan AD, Bidwell LC. Edible cannabis for chronic low back pain: associations with pain, mood, and intoxication. Front Pharmacol. 2024 Sep 24;15:1464005. doi: 10.3389/fphar.2024.1464005. eCollection 2024. PMID 39380911
- See also: CUChange Lab, University of Colorado, Boulder — https://www.colorado.edu/changelab/research

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note: 268 participants were consented for the study. Among those, 253 submitted photos of their experimental product and were thus assigned to product groups. It is not possible to "group" the 15 participants lost to attrition at that point in the study flow.
Groups:
- THC Group: Participants used THC dominant products
- CBD Group: Participants used CBD dominant products
- THC+CBD Group: Participants used products with roughly equivalent proportions of THC and CBD
Period: Overall Study
Arm/Group | THC Group | CBD Group | THC+CBD Group
Started | 38 | 97 | 118
Completed | 36 | 96 | 117
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | THC Group | CBD Group | THC+CBD Group | Total
Number analyzed (Participants) | 36 | 96 | 117 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.92 (15.02) | 50.18 (14.49) | 46.06 (16.38) | 46.3 (16.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 15 | 58 | 68 | 141
  Male | 20 | 37 | 47 | 104
  Transgender/non-binary | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 11 | 17
  Not Hispanic or Latino | 33 | 92 | 105 | 230
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 36 | 96 | 117 | 249
Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Participants' current pain intensity was measured via a single item from the Pain Intensity Short Form 3a which asked, "What is your level of lower back pain currently?" and was rated on a scale of 0 = "no pain" to 10 = "worst imaginable pain"
  units on a scale | 3.2 (0.93) | 3.37 (0.92) | 3.45 (0.97) | 3.4 (0.94)

OUTCOME MEASURES:

1. Primary Outcome: Pain Interference: Roland Morris Disability Questionnaire (RMDQ)
Description: The Roland Morris Disability Questionnaire assesses self-rated physical disability caused by low back pain. Scores range from 0 to 24, with higher scores indicating more pain interference.
Time Frame: Change over two time points over 2 weeks: Baseline (before 2 weeks of edible use), Pre-Administration (after 2 weeks of use and before acute administration) using the total RMDQ score (0-24).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
score on a scale
  Baseline Pain Interference | 8.028 (3.582) | 9.635 (4.98) | 9.034 (4.495)
  Pain Interference at 2 Weeks | 6.194 (4.407) | 8.031 (5.428) | 7.419 (4.796)

2. Primary Outcome: Inflammation: Circulating Levels of Cytokines
Description: Tests levels of recent inflammation (panel of inflammatory markers) before and after cannabis use. Higher numbers indicate higher levels of circulating pro-inflammatory cytokines. Results are in pg/mL and are separated by the three cytokines: IL-1b, IL-6, and IL-10.
Time Frame: Change over two time points over 2 weeks: Baseline (before 2 weeks of edible use) and Pre-Administration (after 2 weeks of use and before acute administration).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 25 | 79 | 96
pg/mL
  Baseline IL-1b blood levels | 6.685 (9.261) | 8.422 (13.766) | 7.829 (11.214)
  IL-1b Blood Levels at 2 Weeks | 6.816 (9.138) | 8.031 (13.274) | 8.014 (11.831)
  Baseline IL-6 Blood Levels | 3.071 (2.769) | 3.994 (4.438) | 3.538 (3.538)
  IL-6 Blood Levels at 2 Weeks | 3.101 (3.091) | 3.639 (4.542) | 3.168 (2.979)
  Baseline IL-10 Blood Levels | 6.183 (8.65) | 7.362 (12.256) | 8.565 (13.513)
  IL-10 Blood Levels at 2 Weeks | 6.184 (8.546) | 7.007 (12.337) | 8.563 (13.842)

3. Primary Outcome: Flanker Inhibitory Control Attention Task (FICA) & International Shopping List Task (ISLT)
Description: Co-outcomes testing cognitive impairment in the domains of immediate and delayed recall (ISLT) and attention and inhibitory control (FICA). Cognitive outcomes are measured in standard scores (e.g. Range of >70 to >140 (Mean of 100 and SD of 15) with higher scores indicating better performance) and can be averaged to reflect a Standard score of overall cognitive function.
Time Frame: Change over two time points over 2 weeks: Baseline (before 2 weeks of edible use), Pre-Administration (after 2 weeks of use and before acute administration).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 93 | 117
score on a scale
  Baseline Flanker Scores | 101.806 (6.528) | 98.606 (7.355) | 99.974 (8.074)
  2 Week Flanker Scores | 102.667 (6.963) | 100.207 (6.657) | 101.063 (8.326)
  Baseline ISLT Scores | 99.886 (14.652) | 98.499 (12.514) | 102.37 (16.359)
  2 Week ISLT Scores | 99.756 (16.278) | 98.325 (13.744) | 100.321 (16.206)

4. Primary Outcome: Functional Assessment of Cancer Therapy Cognitive Scale (FACT-Cog)
Description: Subjective report of cognitive function using the Perceived Cognitive Impairments subscale of the Functional Assessment of Cancer Therapy Cognitive Scale (FACT-Cog). Possible scores range from 0-80 where higher scores are associated with higher levels of perceived impairment.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
score on a scale
  Baseline Perceived Impairments Rating | 15.528 (11.388) | 14.14 (11.834) | 13.978 (11.226)
  2 Week Perceived Impairments Rating | 12.52 (9.913) | 14.037 (12.77) | 12.743 (10.155)

5. Secondary Outcome: Pain Intensity: Current Pain Using NIH Pain Intensity Scale.
Description: Test effects of cannabinoids on pain using the NIH Pain intensity scale for "current pain" (on a scale from 0-10 with 10 being the worst).
Time Frame: Change over 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
score on a scale
  Baseline Pain Intensity Rating | 2.2 (0.933) | 2.366 (0.918) | 2.448 (0.972)
  2-Week Pain Intensity Rating | 3.091 (1.792) | 3.204 (1.948) | 3.288 (2.064)

6. Secondary Outcome: Health & Wellbeing
Description: Self-report measure across primary domains of diet, assessment of sleep quality, and health-related well-being. Each domain was assessed with the following single items:
  Diet: "In general, how healthy is your overall diet? Would you say" (response options 0- excellent; 1- very good; 2- good; 3- fair; 4- poor) Sleep Quality: "During the past 2 weeks, how would you rate your sleep quality overall?" (response options 0- very good; 1- fairly good; 2- fairly bad; 3- very bad") Health Related Wellbeing: "In general, how would you describe your health?" (response options 0- excellent; 1- very good; 2- good; 3- fair; 4- poor)
Time Frame: Change over 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
units on a scale
  Baseline Self Reported Diet | 1.58 (0.94) | 1.56 (0.96) | 1.44 (0.92)
  2 Week Self Reported Diet | 1.54 (0.90) | 1.64 (0.82) | 1.50 (0.96)
  Baseline Sleep Quality | 1.31 (0.79) | 1.27 (0.72) | 1.22 (0.67)
  2 Week Sleep Quality | 1.00 (0.66) | 1.19 (0.63) | 1.06 (0.61)
  Baseline Health-Related Wellbeing | 1.58 (0.84) | 1.52 (0.88) | 1.39 (0.79)
  2 Week Health-Related Wellbeing | 1.44 (0.95) | 1.55 (0.83) | 1.49 (0.76)

7. Secondary Outcome: Pittsburgh Sleep Quality Assessment (PSQI)
Description: The Pittsburgh Sleep Quality Assessment (PSQI) is a self-report assessment of sleep quality.9 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances (Scores range from 0 to 21 overall, with scores greater than 5 suggesting significant sleep difficulties).
Time Frame: Change over 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
score on a scale
  Baseline PSQI Scores | 8.22 (3.54) | 8.39 (3.67) | 7.46 (3.87)
  4 Week PSQI Scores | 5.85 (3.09) | 7.07 (3.74) | 6.14 (3.42)

8. Secondary Outcome: Motor Function
Description: Motor control assessed via dynamic sway and proprioception. Motor outcomes were aggregated to reflect a Z-score of overall motor function. Scores reported below are sum of Motor Battery Balance z-scores (Eyes Open, Eyes Closed, and Head Back). Higher scores correspond to worse balance- there is not a maximum score.
Time Frame: Change over 2 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 32 | 93 | 109
z-score
  Baseline z-score | 0.019 (0.006) | 0.023 (0.013) | 0.021 (0.007)
  2 Week z-score | 0.018 (0.006) | 0.023 (0.011) | 0.02 (0.006)

9. Secondary Outcome: Depression and Stress
Description: The DASS21 is a 21-item scale that measures self-reported change in anxiety, depression, and stress symptoms. Participants are asked to use 4-point severity/frequency scales (higher values indicate greater severity) to rate the extent to which they have experienced each state. For this aim, the Depression and Stress subscales were used.
  Depression subscale score range 0-21 Normal (0 to 4), Mild (5 to 6), Moderate, (7 to 10), Severe (11 to 13), Extremely Severe (14 and above) Stress subscale score range 0-33 Normal (0 to 14), Mild (15 to 18), Moderate, (19 to 25), Severe (26 to 33)
Time Frame: Change over 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
score on a scale
  Baseline Depression score | 7.111 (6.369) | 6.188 (7.41) | 6.872 (8.197)
  2 Week Depression Score | 5.939 (7.132) | 5.532 (6.508) | 5.856 (7.364)
  Baseline Stress Score | 9.667 (7.716) | 9.417 (8.135) | 10.068 (7.991)
  2 Week Stress Score | 8.545 (7.023) | 8.596 (8.042) | 8.198 (6.959)

10. Secondary Outcome: Acute Cognitive Impairment: Flanker Inhibitory Control Attention Task (FICA) and International Shopping List Task (ISLT).
Description: Co-outcomes testing cognitive impairment after acute use of cannabis in the domains of immediate and delayed recall (ISLT) and and attention and inhibitory control (FICA). Cognitive outcomes are measured in standard scores (e.g. Range of <70 to >140 (Mean of 100 and SD of 15) with higher scores indicating better performance) and can be averaged to reflect a Standard score of overall cognitive function.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: standard score
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 93 | 117
standard score
  Baseline Sum Cognitive Score | 100.619 (8.115) | 98.281 (7.694) | 100.904 (10.296)
  2 Week Sum Cognitive Score | 101.675 (9.226) | 99.615 (8.166) | 100.91 (9.944)

11. Secondary Outcome: Patient Global Impression of Change: Global Impression of Change Scale (PGIC).
Description: Patient Global Impression of Change Scale (PGIC) measures self-reported change on a 1-7 scale (i.e. from 1 (very much worse) to 7 (very much improved) in pain. Changes in this measure will be tested in relation to THC and CBD blood levels. Scale possible score range 1-7, with higher scores indicating the largest amount of possible change. Importantly, it is a subjective self-assessment of change and is only measured at the 2 week timepoint.
Time Frame: Change over 2 week primary exposure period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 33 | 94 | 111
score on a scale | 4.97 (0.847) | 4.745 (0.867) | 4.856 (0.862)

12. Other Pre Specified Outcome: Exploratory: Daily Follow-up Messages
Description: Brief self-report from participants on pain and sleep in the past 24 hours. These are 1-item novel questions in a daily, text based survey. Pain and sleep are on a scale of 1-10, with higher numbers being more pain or better sleep. Score is an average rating over 14 days.
Time Frame: 2 weeks (daily)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 116
units on a scale
  Pain Rating | 2.989 (1.848) | 3.247 (2.033) | 3.322 (2.083)
  Sleep Rating | 5.426 (1.823) | 4.916 (1.657) | 5.193 (1.801)

13. Other Pre Specified Outcome: Exploratory: Monthly Follow-up Surveys
Description: Self-report from participants on pain levels (0-10 with 10 being worst pain), sleep quality (0-10 with 10 being best sleep), perceived cognitive ability (0 - 27 with 27 being the best), perceived cognitive impairments (0-72 with 72 being the worst), and general health (0-4 with 4 being best). Scores are reported as average scores reported once a month over six months.
Time Frame: 6 months (monthly)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 33 | 89 | 105
units on a scale
  Monthly Pain Rating | 3.067 (3.15) | 2.844 (2.974) | 3.216 (3.153)
  Monthly Sleep Quality | 5.763 (1.79) | 5.837 (1.708) | 5.595 (1.626)
  Monthly Perceived Cognitive Ability | 18.78 (6.152) | 19.408 (6.134) | 18.473 (6.612)
  Monthly Perceived Cognitive Impairments | 5.756 (10.222) | 4.88 (7.918) | 7.718 (14.185)
  Monthly General Health Rating | 1.367 (0.893) | 1.606 (0.745) | 1.588 (0.777)

14. Other Pre Specified Outcome: Objective Physical Activity/Exercise
Description: Physical activity via objective daily data on wearable watch as measured by average minutes of moderate to vigorous physical activity (MVPA).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 31 | 82 | 94
minutes | 1610.258 (773.122) | 1830.455 (1103.797) | 1723.745 (1081.798)

15. Other Pre Specified Outcome: Physical Activity/Exercise
Description: Physical activity via subjective self-report data using the Stanford Leisure-Time Activity Categorical item with 6 item responses (L-CAT; 1-6). Scores are reported as a mean between 1 and 6, larger numbers correspond to higher levels of activity.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 36 | 96 | 117
score on a scale
  Baseline Physical Activity | 3.806 (1.39) | 3.417 (1.202) | 3.573 (1.328)
  2 Week Physical Activity | 3.788 (1.293) | 3.277 (1.177) | 3.279 (1.097)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: This study was quasi-observational and minimally invasive.
Arm/Group | THC Group | CBD Group | THC+CBD Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/95 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/95 | 0/117
Other Adverse Events (participants affected / at risk) | 0/36 | 0/95 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT03522324/Prot_SAP_000.pdf